CLINICAL TRIAL: NCT04918264
Title: Fluoropyrimidine Tailored-dose Based on Uracil Concentration in Patients Treated for Digestive Carcinomas: Evaluation of Clinical Practice
Acronym: URACILMPACT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0489
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Digestive Carcinoma
Keywords: Uracil; DPYD; Toxicity; Clinical practice; Overall survival
MeSH Terms: interventions — Fluorouracil; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uracil concentration <16 ng/mL: Patients were included in this arm if they have digestive cancer and an uracil dosage <16 ng/mL performed between February 2018 to January 2020, and if they received at least one cycle of fluoropyrimidine-based chemotherapy in one of the four oncology departments (Hopital Edouard Heriot [Lyon], Centre Hospitalier de Lyon Sud [Lyon], Hopital de la Croix Rousse [Lyon].
  Interventions: Drug: Fluoropyrimidine treatment (5-FU or capecitabine) and dosage; Other: Uracil dosage; Behavioral: Overall survival
- Uracil concentration ≥16 ng/mL: Patients were included in this arm if they have digestive cancer and an uracil dosage <16 ng/mL performed between February 2018 to January 2020, and if they received at least one cycle of fluoropyrimidine-based chemotherapy in one of the four oncology departments (Hopital Edouard Heriot [Lyon], Centre Hospitalier de Lyon Sud [Lyon], Hopital de la Croix Rousse [Lyon].
  Interventions: Drug: Fluoropyrimidine treatment (5-FU or capecitabine) and dosage; Other: Uracil dosage; Behavioral: Overall survival

INTERVENTIONS:
Drug: Fluoropyrimidine treatment (5-FU or capecitabine) and dosage — In each group with an uracil dosage; at cycle 1; capecitabine or continuous 5-FU dose percentage will be evaluate retrospectively in our database
Other: Uracil dosage — For each patient, uracil concentration will be evaluate and patients will be compared based on 16 ng/mL as threshold.
Behavioral: Overall survival — For each group of patient, on 16 ng/mL as threshold for uracil concentration, overall survival will be compared betwen the two groups of patients (Uracil <16 vs Uracil ≥16).

SUMMARY:
Digestive carcinomas chemotherapies regimen are mostly based on fluoropyrimidine drugs (5-Fluorouracil (5-FU) or capecitabine). 5-FU is mainly catabolised by dihydropyrimidine dehydrogenase (DPD) and partial or complete DPD deficiency can cause severe adverse reactions. Different strategies have been proposed to predict DPD deficiency; the two main approaches are phenotyping the enzyme activity (directly or indirectly), or genotyping the four main polymorphisms associated with 5-FU-toxicity. In February 2018, the French medicines agency (Agence nationale de sécurité du médicament et des produits de santé, ANSM) recommended DPD genotyping for all patients receiving fluoropyrimidine-based treatment to improve its safety as compared to the European Medicines Agency (EMA)13 and others pharmacogenetics working group.

In December 2018, a new guideline from the French cancer institute (Institut National Du Cancer, INCa) and the French health authority (Haute Autorité de Santé, HAS) recommended the measurement of the uracil blood level before genotyping DPD and dose adaptation if this level is greater than 16 ng/mL. The aim herein is to assess how this recommendation has been implemented in clinical routine. 5-FU displays a dose-response relationship regarding both its efficacy and its toxicity, did tailored-dose impair the treatment efficacy as it decreased the risk of toxicity? To address that matter we conducted a retrospective study to evaluate how fluoropyrimidine dosage is adapted to uracil concentration with an emphasis on how patients outcome were affected. We compared time to failure and overall survival between patients with an uracil concentration < 16 ng/mL and > or = 16 ng/mL.

ELIGIBILITY:
Inclusion Criteria:

* Digestive cancer
* An uracil dosage performed between February 2018 to January 2020
* Received at least one cycle of fluoropyrimidine-based chemotherapy in one of the three oncology departments (Hopital Edouard Heriot [Lyon], Centre Hospitalier de Lyon Sud [Lyon], Hopital de la Croix Rousse [Lyon]).

Exclusion Criteria:

* Age limit less than 18 years
* Not treated with fluoropyrimidine based chemotherapy
* Missing data for uracil concentration or chemotherapy dosage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included in this retrospective study if they have digestive cancer and an uracil dosage performed between February 2018 to January 2020, and if they received at least one cycle of fluoropyrimidine-based chemotherapy in one of the three oncology departments (Hopital Edouard Heriot [Lyon], Centre Hospitalier de Lyon Sud [Lyon], Hopital de la Croix Rousse [Lyon]. The following characteristics will be review: histology, stage (localized vs metastatic disease), chemotherapy regimen, dose percentage of fluoropyrimidine, fluoropyrimidine induced-toxicity, time to failure and overall survival.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Overall survival according to plasma uracil concentration | Last completion date March 30th 2021

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Edouard Heriot, Centre Hospitalier de Lyon Sud [Lyon], Hopital de la Croix Rousse [Lyon], Lyon
  - Hopital de la Croix Rousse, Lyon
  - Centre Hospitalier de Lyon Sud, Pierre-Bénite